CLINICAL TRIAL: NCT01060865
Title: Treatment of Essential Hypertension With Rasilez. Evaluation of Different Methods of Blood Pressure Measurements - Efficacy and Safety Evaluation
Brief Title: Evaluation of Aliskiren Efficacy by Different Methods of Blood Pressure Measurements
Acronym: REALITY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The participants signed an old version of the informed consent.
Sponsor: Meir Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100AIL02T
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2011-05

CONDITIONS: Blood Pressure, High
Keywords: hypertension; aliskiren; Blood Pressure Monitoring, Ambulatory
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aliskiren (Experimental): only one arm with the experimental drug [aliskiren]
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — 150 mg during the first two weeks , 300 mg for another 10 weeks
  Other Names: Blood Pressure; Ambulatory Blood Pressure monitor; Self measured home blood pressure

SUMMARY:
Almost 50% of hypertensive patients remain uncontrolled. Clinical decisions are mostly based on office blood pressure,despite the fallacies of this method of measurement. Other reasons for not achieving blood pressure targets are lack of 24-hr efficacy and tolerability of existing anti-hypertensive drug classes. Aliskiren (Rasilez®) is a new antihypertensive drug, given once a day.

The purpose of the REALITY study-[tREAtment of essentiaL hypertension with rasIlez. evaluation of different methods of blood pressure measurements - efficacy and safeTY evaluation -] is to evaluate the efficacy, and tolerability of aliskiren in a "real life" setting. The efficacy of the drug will be evaluated using 24 hour ambulatory blood pressure monitoring (ABPM). Results will be compared with office, nurse or self blood pressure monitoring. This comparison will allow to decide which follow-up technique is better for those hypertensive patients.

DETAILED DESCRIPTION:
This is a single centre observational uncontrolled prospective study, Hypertensive patients that are either treatment naïve or uncontrolled on current monotherapy and meet all inclusion and exclusion criteria, will be assigned to Rasilez treatment (start for 2 weeks on 150 mg and if well tolerated the dosage will be increased to 300 mg). The treatment will then be continued for additional 10 weeks. Rasilez can be administrated as monotherapy or as add on to other antihypertensive (patients currently on single medication).

The patient will have additional visits at week 6, and at week 12 For all eligible patients a 24 h ABPM test will be performed at the week prior to visit 2 (treatment initiation) and at the week prior to the final visit.

Each patient will receive an automatic blood pressure monitor [OMRON MX3 plus] for SBPM measurements, The monitor will be provided by the sponsor for the whole study period. The patient will be trained for blood pressure measurements. SBPM will be performed twice a week [morning and evening] Nurse blood pressure measurements will be performed at each visit, after 10 minutes of rest, prior to the medical visit.

Office blood pressure will be performed by the physician at each visit Blood samples for electrolytes, renal function, liver function and hematology, will be taken at base line visit, at week 2 and at week 12 Other antihypertensive can be added at any time during the study, according to the decision of the investigator, except ACE inhibitors and ARBs.

AEs have to be reported at the appropriate site on the CRF page. In case of discontinuation of aliskiren or interruption of aliskiren treatment the reason has to be given. Serious adverse events (SAEs) have to be documented additionally on the separate SAE form and have to be reported within 24h to the NOVARTIS Pharma, Drug safety department Adherence to treatment will be evaluated using standard formulas. Estimated time for recruitment of 50 patients: One year. Study design scheme Visit 1 -[week -2] physician and nurse BP. Sign inform consent- command ABPM a week prior to visit 2 - SBPM training Visit 2 [week 0] physician and nurse BP. Start Rasilez 150 mg and command laboratory exams prior to next visit.

Visit 3 [week 2] physician and nurse BP. Titrate Rasilez to 300 mg Visit 4 (week 6). physician and nurse BP. ABPM and command lab exams (a week prior to visit 5) Visit 5 (12 weeks) physician and nurse BP SBPM data will be collected at visit 2,3,4 and 5.

Efficacy will be defined in terms of therapeutic goals expressed as target blood pressures according to WHO and ESH [ for SBPM and ABPM] criteria:

Office Blood Pressure: Diastolic blood pressure (DBP) ≤ 90 mmHg and Systolic blood pressure (SBP) ≤ 140 mmHg for non-diabetics or DBP≤ 80 mmHg and SBP≤ 130 mmHg for diabetics, respectively.

SBPM : DBP ≤ 85 mmHg and SBP ≤ 135 mmHg 24 h ABPM: DBP≤ 130/80 mmHg SBP≤ 130 mmHg, Awake DBP ≤ 85 mmHg, Awake SBP ≤ 135 mmHg Asleep DBP ≤70 mmHg, asleep SBP ≤ 70 mmHg. Effectiveness and Safety will also be evaluated taking into consideration patient compliance

Safety assessments:

Safety will be assessed by means of (S)AE reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension at visit 1 defined as office blood pressure <140/90 mmHg and a 24 h ABPM >130/80 mmHg with a day time BP (extracted from the 24h ABPM) >135/85 mmHg
2. Male and female
3. Age 18-80
4. Every patient that in the medical opinion of the treating physician is eligible for Rasilez treatment
5. Willing to sign an informed consent

Exclusion Criteria:

1. Use of more then 1 anti hypertensive medication at visit 1 (fixed combination is considered as two drugs)
2. Use of ACEI or ARB at base line visit
3. Pregnant women
4. WOCB - (will follow the usual limitations)
5. Use of certain medications (e.g. Cyclosporine, Verapamil, Quinidine)
6. Uncontrolled DM (investigator decision)
7. Any of the following in the last six months: MI, Stroke, CABG, PTCI
8. Congestive HF requiring pharmacological treatment
9. Renal Failure, defined as serum creatinine equal or great than 1.5 mg% [confirmed twice] or hyperkalemia defined as serum potassium equal or great that 5 meq/l [confirmed twice]
10. Malignancy that required Chemotherapy in the last 3 years
11. Any medical or none medical condition that in the eyes of the investigator will not allow the patient to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with controlled blood pressure with office BP measurements, nurse measurements and SBPM, from baseline to week 12, compared and ABPM. | 12 weeks

SECONDARY OUTCOMES:
Compare the SBP/DBP lowering efficacy of Rasilez treatment in patients with essential hypertension as measured by 4 different methods - 24h Ambulatory BP measurement, Office BP, Home BP and Nurse BP measurement. | 12 weeks
To assess patient adherence to treatment. | 2, 6 and 12 weeks
To evaluate the safety profile of Rasilez treatment in patients with essential hypertension. | 2, 6 and 12 weeks
Evaluate the antihypertensive effect of Rasilez in "real life", based on the 24h ABPM changes from base line to week 12. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Podjarny, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit health services, Herzliya, Hasharon Area, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schmieder RE, Philipp T, Guerediaga J, Gorostidi M, Bush C, Keefe DL. Aliskiren-based therapy lowers blood pressure more effectively than hydrochlorothiazide-based therapy in obese patients with hypertension: sub-analysis of a 52-week, randomized, double-blind trial. J Hypertens. 2009 Jul;27(7):1493-501. doi: 10.1097/HJH.0b013e32832be593. PMID 19444142
- [Background] Gradman AH, Schmieder RE, Lins RL, Nussberger J, Chiang Y, Bedigian MP. Aliskiren, a novel orally effective renin inhibitor, provides dose-dependent antihypertensive efficacy and placebo-like tolerability in hypertensive patients. Circulation. 2005 Mar 1;111(8):1012-8. doi: 10.1161/01.CIR.0000156466.02908.ED. Epub 2005 Feb 21. PMID 15723979
- [Background] Uresin Y, Taylor AA, Kilo C, Tschope D, Santonastaso M, Ibram G, Fang H, Satlin A. Efficacy and safety of the direct renin inhibitor aliskiren and ramipril alone or in combination in patients with diabetes and hypertension. J Renin Angiotensin Aldosterone Syst. 2007 Dec;8(4):190-8. doi: 10.3317/jraas.2007.028. PMID 18205098
- [Background] Verdecchia P, Calvo C, Mockel V, Keeling L, Satlin A. Safety and efficacy of the oral direct renin inhibitor aliskiren in elderly patients with hypertension. Blood Press. 2007;16(6):381-91. doi: 10.1080/08037050701717014. PMID 18058456
- [Background] Jordan J, Engeli S, Boye SW, Le Breton S, Keefe DL. Direct Renin inhibition with aliskiren in obese patients with arterial hypertension. Hypertension. 2007 May;49(5):1047-55. doi: 10.1161/HYPERTENSIONAHA.106.084301. Epub 2007 Mar 12. PMID 17353513
- [Background] Burt VL, Cutler JA, Higgins M, Horan MJ, Labarthe D, Whelton P, Brown C, Roccella EJ. Trends in the prevalence, awareness, treatment, and control of hypertension in the adult US population. Data from the health examination surveys, 1960 to 1991. Hypertension. 1995 Jul;26(1):60-9. doi: 10.1161/01.hyp.26.1.60. PMID 7607734
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Background] Dolan E, Stanton AV, Thom S, Caulfield M, Atkins N, McInnes G, Collier D, Dicker P, O'Brien E; ASCOT Investigators. Ambulatory blood pressure monitoring predicts cardiovascular events in treated hypertensive patients--an Anglo-Scandinavian cardiac outcomes trial substudy. J Hypertens. 2009 Apr;27(4):876-85. doi: 10.1097/HJH.0b013e328322cd62. PMID 19516185